CLINICAL TRIAL: NCT03422016
Title: The Incidence of Altered Light Responses in Children With Autistic Spectrum Disorders
Brief Title: Electroretinogram in Autistic Spectrum Disorders
Acronym: ERG in ASD
Status: Completed | Type: Observational
Sponsor: Great Ormond Street Hospital for Children NHS Foundation Trust (Other)
Collaborators: Flinders University (Other); Yale University (Other); Swinburne University of Technology (Other)
Responsible Party: Sponsor
Other Study IDs: 17PP33
Record Dates: First submitted 2018-01-30; First posted 2018-02-05 (Actual); Last update posted 2022-01-11 (Actual); Status verified 2022-01

CONDITIONS: Autism Spectrum Disorder
Keywords: electroretinogram
MeSH Terms: conditions — Autism Spectrum Disorder | interventions — Electroretinography

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- autistic spectrum disorder: intelligence quotient IQ>85 age 4-25yrs
  Interventions: Diagnostic Test: electroretinogram (ERG)
- control: age 4-25yrs no eye disorder
  Interventions: Diagnostic Test: electroretinogram (ERG)

INTERVENTIONS:
Diagnostic Test: electroretinogram (ERG) — an ERG is a measure of the eyes response to a flash of light

SUMMARY:
This study aims to find out the incidence of a reduced light adapted electroretinogram (ERG) b-wave amplitude in children with a diagnosis of Autism Spectrum Disorders (ASD).

DETAILED DESCRIPTION:
Autism Spectrum Disorder (ASD) is a neurodevelopmental condition which becomes apparent as children grow. Children with ASD are slow to develop language and have problems interacting socially with others. It is not clear why ASD occurs, but there is some evidence that the signals that tell the brain how to grow are altered which causes the brain to develop and function differently in people with ASD. Eyes develop from the same embryonic tissue as the brain. This means that the retina, which is the light sensitive layer at the back of the eye, shares the same signals as the brain. Investigators can listen to retinal signals outside the eye and the retina can, in this way, act as an accessible part of the brain.

The investigators will detect retinal signals as electrical messages. Sensors placed near the eye pick up the electrical changes in the retina each time a light flashes. This non-invasive, routine clinical test is called an electroretinogram, (ERG). The investigators have carried out a study that showed differences in the ERGs recorded from adults with ASD compared to control participants.

The main aim of this project is find out how common ERG differences are in children with ASD compared to controls. If it is common, investigators could use the ERG to make an earlier diagnosis of ASD and help families sooner. It could help investigators better understand the way the ASD brain signals and give investigators a way of measuring if therapies work.

ELIGIBILITY:
Inclusion Criteria:

* cohort 1: individuals with diagnosis ASD with an IQ measure exceeding 85
* cohort 2: typically developed controls without diagnosis of ASD

Exclusion Criteria:

* a history of eye disease or treatment or seizure medicines that may alter retinal function

Ages: 4 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: individuals diagnosed with ASD and typically developing controls
Sampling Method: Non-Probability Sample
Enrollment: 177 (Actual)
Dates: Start 2018-09-03 (Actual); Primary Completion 2020-03-03 (Actual); Study Completion 2020-04-03 (Actual)

PRIMARY OUTCOMES:
light adapted electroretinogram | 12 months
  incidence of reduced light adapted electroretinogram in children with a diagnosis of autism spectrum disorder

CONTACTS AND LOCATIONS:
Overall Officials: Dorothy A Thompson, PhD, Principal Investigator — Consultant Clinical Scientist Visual Electrophysiology, Great Ormond Street Hospital for Children London UK; Paul Constable, PhD, Study Director — Head Of Teaching Optometry, Flinders Vision Autism Centre, Flinders University, Australia; James McPartland, PhD, Principal Investigator — Associate Professor of Child Psychiatry and Psychology, Director, Yale Developmental Disabilities Clinic, Yale University, USA
Locations (4):
- Yale University, New Haven, Connecticut, United States
- Australia (2):
  - Flinders University, Adelaide, South Australia
  - Swinburne University of Technology, Melbourne
- Great Ormond Street Hospital for Children NHS Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No